CLINICAL TRIAL: NCT07046208
Title: Effects os Physiotherapeutic Rehabilitation on Cardiovascular Autonomic Modulation and Biomarkers Inflammatory and Cardiac Conditions in Patients With Long Covid
Brief Title: Effects os Physiotherapeutic Rehabilitation on Function Autonomic and Inflammatory in Patients With Long Covid
Acronym: LongCovidRehab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Luiz Fábio Magno Falcão, PhD, Researcher, Universidade do Estado do Pará
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 36459920400005174; 4252664 (Registry Identifier: Comitê de ética em pesquisa da Universidade do Estado do Pará)
Record Dates: First submitted 2025-06-29; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Long COVID; Heart Rate Variability (HRV); Cardiac Biomarkers; Inflammatory Biomarkers
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation for long covid (Experimental): Physioterapy protocol
  Interventions: Other: physiothreapy protocol

INTERVENTIONS:
Other: physiothreapy protocol — Aerobic training (treadmill or exercise bike) for 15 minutes, anaerobic training at the weight training station, performing exercises for the upper limbs (bench press and front pull) and lower limbs (180º leg press and extension chair) with weight determined by the 1 Repetition Maximum (1RM) test, performing 3 sets of 12-15 repetitions (depending on the session) and respiratory muscle training using POWERbreathe (30-40% of the MIP performed in the manovacuometry test).

SUMMARY:
Introduction: Long COVID is characterized by persistent symptoms that persist for weeks or months after the acute phase of infection, with a significant impact on the cardiovascular and autonomic systems. Objectives: This study aims to evaluate the effects of a physiotherapeutic rehabilitation protocol on cardiovascular autonomic modulation and on inflammatory and cardiac biomarkers in patients with Long COVID. Methodology: This is a controlled clinical trial, carried out in a cardiorespiratory rehabilitation outpatient clinic, involving individuals with a clinical diagnosis of Long COVID undergoing a protocol of 20 aerobic, anaerobic and respiratory rehabilitation sessions. Heart rate variability (HRV) variables will be analyzed using linear and non-linear methods, in addition to serum levels of CKMB, LDH, ferritin and C-reactive protein. Expected results: Rehabilitation is expected to provide an improvement in autonomic function and a reduction in inflammatory and cardiac markers, contributing to the understanding of the pathophysiological mechanisms of Long COVID and helping to propose evidence-based therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* aged 20 and 59 years
* clinical evaluation and undergoing clinical follow-up of Post COVID-19.
* least one persistent COVID-19-related symptom.

Exclusion Criteria:

* incomplete data.
* presence of a pacemaker
* use of antihypertensive drugs that alter HRV
* persistent pulmonary alterations
* persistent desaturation
* anaemia or presence of reinfection.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Autonomic Modulation | Before and afther the intervention 3 months.
  cardiofrequency meter

SECONDARY OUTCOMES:
Inflammation | Before and the afther 3 months
  the cardiac and inflammatory biomarkers, creatine phosphokinase isoenzyme MB (CKMB) associated with lactate dehydrogenase (LDH) and ferritin can be analysed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marques KC, Silva CC, Trindade SDS, Santos MCS, Rocha RSB, Vasconcelos PFDC, Quaresma JAS, Falcao LFM. Reduction of Cardiac Autonomic Modulation and Increased Sympathetic Activity by Heart Rate Variability in Patients With Long COVID. Front Cardiovasc Med. 2022 Apr 29;9:862001. doi: 10.3389/fcvm.2022.862001. eCollection 2022. PMID 35571200

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT07046208/Prot_SAP_ICF_000.pdf